CLINICAL TRIAL: NCT00427401
Title: A Double Blind, Placebo Controlled, Parallel Group Study To Evaluate The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of PF-00915275 After Oral Administration To Subjects With Type 2 Diabetes Mellitus For 4-Weeks
Brief Title: A Study To Evaluate PF-00915275 In Subjects With Type 2 Diabetes Mellitus For 4-Weeks
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated May 7, 2007. The study stopped due to tablet formulation issues. No safety issues were involved in the termination decision.
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A8441003
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: PF-00915275

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of PF-00915275 following administration to adult human subjects with T2DM for 4-weeks. The primary end point is glucose lowering (24 hour mean glucose concentration).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* HbA1c > 7.5%.

Exclusion Criteria:

* Recent (within the past 12 months) evidence or history of unstable concomitant disease.
* Treatment with any oral hypoglycemic agent within 3 months before enrollment.
* The exception to these criteria is that subjects who are currently taking metformin hydrochloride, in a stable dose (that is no changes in dose) for treatment of their diabetes within the past 3 months or longer of enrollment may participate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2007-02; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary end point is glucose lowering (24 hour mean glucose concentration).

SECONDARY OUTCOMES:
Fasting blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8441003&StudyName=A%20Study%20To%20Evaluate%20PF-00915275%20In%20Subjects%20With%20Type%202%20Diabetes%20Mellitus%20For%204-Weeks%20